CLINICAL TRIAL: NCT05831709
Title: De Invloed Van Hormoonsubstitutietherapie en Gesuperviseerde Training op Lichaamssamenstelling, Cardiovasculair Risico en Insulinegevoeligheid Bij Postmenopauzale Vrouwen
Brief Title: The Influence of Hormone Replacement Therapy and Supervised Exercise Training on Body Composition, Cardiovascular Risk and Insulin Sensitivity in Postmenopausal Women
Acronym: OPERATE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ONZ-2023-0015
Record Dates: First submitted 2023-04-12; First posted 2023-04-26 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Postmenopause; Menopausal Complaints
MeSH Terms: interventions — Resistance Training

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Supervised training + immediate hormone substitution therapy per SOC (Experimental)
  Interventions: Other: Exercise program; Drug: Hormonal substitution therapy per SOC
- Supervised training + delayed hormone substitution therapy per SOC (Experimental)
  Interventions: Other: Exercise program
- Delayed supervised training + immediate hormone substitution therapy per SOC (Active Comparator)
  Interventions: Drug: Hormonal substitution therapy per SOC
- Supervised training (Experimental): Subjects who will start hormone substitution therapy in standard of care can participate in the trial and have 50% chance to be randomised in the exercise group.
  Interventions: Other: Exercise program
- No supervised training (No Intervention): Subjects who will start hormone substitution therapy in standard of care can participate in the trial and have 50% chance to be randomised in the non-exercise group.
- Control group (No Intervention): Subjects with menopausal complaints who do not want hormone substitution therapy or supervised training, can also participate in the trial.

INTERVENTIONS:
Other: Exercise program — The intervention consists of a supervised exercise program
  Arms: Supervised training; Supervised training + delayed hormone substitution therapy per SOC; Supervised training + immediate hormone substitution therapy per SOC
Drug: Hormonal substitution therapy per SOC — Subjects take hormonal substitution therapy per standard of care
  Arms: Delayed supervised training + immediate hormone substitution therapy per SOC; Supervised training + immediate hormone substitution therapy per SOC

SUMMARY:
This trial investigates whether supervised training in combination with hormonal substitution therapy has an impact on body composition, cardiovascular risk, risk for dementia, osteoporosis and insulin sensitivity in postmenopausal women.

DETAILED DESCRIPTION:
270 postmenopausal women will be included. Each woman will perform a 12 to 24 weeks sports program with supervised training exercises.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women (diagnosed by physician) with complaints due to menopause
* Indication for hormonal substitution therapy (except for the control group)
* Good general health
* BMI: 20-30 kg/m2
* Only the use of cholesterol-, blood pressure- or/and thyroid-regulating medication is permitted

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 390 (Estimated)
Dates: Start 2023-05-12 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the cardiovascular risk | +12 weeks; +24 weeks
  The cardiovascular risk will be estimated by blood- and urine analysis, blood pressure and a AGE (i.e. Advanced Glycation End products)-reader. There are three timepoints of measurement; once at inclusion, once at 12 weeks, and once at 24 weeks.
Evaluation of the insulin sensitivity | +12 weeks, +24 weeks
  The insulin sensitivity will be estimated by blood- and urine analysis and a AGE (i.e. Advanced Glycation End products)-reader. There are three timepoints of measurement; once at inclusion, once at 12 weeks, and once at 24 weeks.

SECONDARY OUTCOMES:
Evaluation of the body composition | +12 weeks; +24 weeks
  The body composition will be measured using bioimpedance technology (Tanita-scale). The body composition will be measured three times; once at inclusion, once at 12 weeks and once at 24 weeks.
Evaluation of the muscle mass | +12 weeks; +24 weeks
  The musle mass will be evaluated by performing a maximal effort test (i.e. cycling test). This test will be performed three times; once at inclusion, once at 12 weeks, and once at 24 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Ghent University Hospital - Women's Clinic, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No